CLINICAL TRIAL: NCT02291718
Title: Comparison of High Iodine Concentration Contrast Material (Isovue 370) vs Standard Protocol (Isovue 300) in Thoracoabdominal Aortic Computed Tomographic Angiography (CTA) for Radiation Dose Reduction
Brief Title: Thoracoabdominal Arortic CTA Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00048275
Record Dates: First submitted 2014-10-23; First posted 2014-11-14 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-01

CONDITIONS: Thoracic Aortic Aneurysm
Keywords: Suspected or confirmed; TAA; Computed tomography angiography; CTA; Contrast agent; Radiation dose; Thoracoabdominal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Aneurysm, Thoracoabdominal | interventions — Iopamidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Isovue 300 75mL (Active Comparator): Isovue 300 75mL injected 120 kVp 250 mAs
  Interventions: Drug: Isovue
- Isovue 370 75mL (Active Comparator): Isovue 370 75mL injected 100 kVp 240 mAs
  Interventions: Drug: Isovue
- Isovue 370 60mL (Active Comparator): Isovue 370 60mL injected 100 kVp 240 mAs
  Interventions: Drug: Isovue

INTERVENTIONS:
Drug: Isovue — iodine contrast

SUMMARY:
The purpose of this study is to compare the contrast agents and imaging techniques used for thoracoabdominal aortic imaging in CT. Imaging parameters and contrast volume are changed and adjusted based on the contrast agent, since contrast agents have varying iodine concentrations. If the contrast iodine concentration is higher, it may be possible to adjust the imaging parameters and lower the overall radiation dose to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracoabdominal aortic (TAA) CTA
* Able to provide informed consent
* Body Mass Index (BMI) equal to or less than 30

Exclusion Criteria:

* Creatinine greater than 2.0
* Allergy to contrast media
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Isovue 300 (75mL): 75mL Isovue 300 injected 120kvp, 250mAs used to obtain CT scan
- Isovue 370 (75mL): 75mL Isovue 370 injected 100 kVp, 250 mAs used for obtaining CT
- Isovue 370 (60mL): 60mL Isovue 370 injected 100 kVp, 240 mAs used to obtain CT
Period: Overall Study
Arm/Group | Isovue 300 (75mL) | Isovue 370 (75mL) | Isovue 370 (60mL)
Started | 50 | 50 | 50
Completed | 50 | 50 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isovue 300 (75mL) | Isovue 370 (75mL) | Isovue 370 (60mL) | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 15 | 14 | 50
  >=65 years | 29 | 35 | 36 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 27 | 65
  Male | 31 | 31 | 23 | 85

OUTCOME MEASURES:

1. Primary Outcome: Radiation Dose
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: mSv
Arm/Group | Isovue 300 75mL | Isovue 370 75mL | Isovue 370 60mL
Number analyzed (Participants) | 50 | 50 | 50
mSv | 35.1 (6.2) | 25.4 (5.3) | 25.5 (7.0)

2. Secondary Outcome: Signal to Noise Ratio
Description: Calculated as the ratio of mean attenuation values divided by the standard deviation of attenuation values gathered using a circular region of interest in the thoracic aorta.
Time Frame: 30 minutes
Population: Hiatus region of each subject group
Measure: Mean (Standard Deviation); unit: Signal-to-Noise Ratio
Arm/Group | Isovue 300 75mL | Isovue 370 75mL | Isovue 370 60mL
Number analyzed (Participants) | 50 | 50 | 50
Signal-to-Noise Ratio | 12.0 (4.8) | 11.8 (3.5) | 13.8 (6.3)

3. Secondary Outcome: Hounsfield Unit Attenuation Values
Description: Grayscale values on CT scans are given as Hounsfield units. These Hounsfield units reflect the attenuation of x-ray beams traversing the aortic lumen. We will use Hounsfield units to assess whether the tool contrast agents achieve similar attenuation characteristics essential for diagnosing aortic abnormalities. We will use circular regions of interest in the thoracic aorta to extract the Hounsfield unit measurements.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: Hounsfield units
Arm/Group | Isovue 300 75mL | Isovue 370 75mL | Isovue 370 60mL
Number analyzed (Participants) | 50 | 50 | 50
Hounsfield units | 289.7 (23.8) | 400.9 (31.1) | 393.9 (28.1)

4. Secondary Outcome: Variation in Contrast for the Entire Vascular System (coV)
Description: The change in contrast was measured at the proximal segment of the aorta and at the Iliac arteries for each subject.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Isovue 300 75mL | Isovue 370 75mL | Isovue 370 60mL
Number analyzed (Participants) | 50 | 50 | 50
unitless | 0.113 (0.073) | 0.124 (0.063) | 0.107 (0.059)

ADVERSE EVENTS:
Arm/Group | Isovue 300 (75mL) | Isovue 370 (75mL) | Isovue 370 (60mL)
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No